CLINICAL TRIAL: NCT06527898
Title: Hypofractionated Radiotherapy Combined with Immunotherapy for Limited-stage Small-cell Lung Cancer: a Phase II Trial
Brief Title: Hypofractionated Radiotherapy Combined with Immunotherapy for Limited-stage Small-cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-ky302
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Small-cell Lung Cancer
Keywords: Hypofraction radiotherapy, Small cell lung cancer, immune checkpoint inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Immunotherapy

STUDY DESIGN:
Intervention Model Description: Hypofractionated radiotherapy combined with immunotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: hypofractionated radiotherapy with immunotherapy — hypofractionated radiotherapy with Adebrelimab consolidation

SUMMARY:
Concurrent chemoradiotherapy has long been the standard modality for locally advanced small-cell lung cancer, which could achieve median overall survival of 25 mos. Conventional fractionation of 66Gy/33f and hyperfractionation of 45Gy/30f twice daily have been acknowledged as the two standard radiotherapy modalities according to CONVERT study. With the introduction of immune checkpoint inhibitors, ADRIATIC study concluded that consolidative Durvalumab after concurrent chemoradiotherapy could achieve a far longer median overall survival of 55.9 months compared with 33.4 months for concurrent chemoradiotherapy. Recently, several studies have demonstrated the safety and efficacy of hypofractionated radiotherapy (3 to 4 Gy) for limited-stage small-cell lung cancer. Hypofractionated radiotherapy processes the advantage of short treatment duration compared with conventional fractionated radiotherapy, which may allow the early participation of immunotherapy. Therefore, we suppose that whether hypofractionated radiotherapy combined with immunotherapy could improve the survival of limited-stage of small-cell lung cancer.

DETAILED DESCRIPTION:
Trial design: To enroll 45 patients diagnosed with limited stage small-cell lung cancer to receive concurrent chemoradiotherapy with consolidative Adebrelimab maintenance.

Primary endpoint: Progression-free Survival Secondary endpoint: 2-year progression-free survival, 2-year overall survival rate.

All enrolled patients are proposed to receive concurrent chemoradiotherapy and consolidative Adebrelimab maintenance up to 2 years. After concurrent chemoradiotherapy, hippocampus-sparing prophylactic cranial irradiation or MRI surveillance are both allowed.

Chemotherapy: Etoposide 80-100mg/m2 day 1, 2, 3 and cisplatin 75-80mg/m2 day 1 & carboplatin AUC 5 day 1 q3w for totally 6 cycles.

Radiotherapy began at the second cycle of chemotherapy followed by hippocampus-sparing prophylactic cranial irradiation or MRI surveillance.

Immunotherapy consolidation began at the third cycle of chemotherapy: Adebrelimab 1200mg q3w to 2 year or disease progression & untolerated toxicity.

Radiotherapy details:

Radiotherapy CT simulation: 4-Dimensional CT (4D-CT) with intravenous contrast is recommended for simulation. Scan thickness should be less than 5 mm. Thermal mask or vacuum bag is recommended.

Target Delineation: Considering hypofraction and involved field irradiation (IFI), only Internal Tumor Volume (ITV) should be delineated without the need to delineate Clinical Tumor Volume (CTV).

Delineation of ITV: ITV should include pulmonary gross tumor and metastatic mediastinal lymph nodes. PET-CT registration with simulation CT is recommended for patients with obstructive atelectasis. For patients with suspected mediastinal lymph nodes, Endobronchial Ultrasound-guided Transbronchial Needle Aspiration (EBUS-TBNA) is recommended.

Production of Planning Tumor Volume (PTV): PTV is produced by a margin of 5 mm added to ITV. Modification of PTV is suggested to respect anatomic boundary.

Dosimetric Limitation: 95% prescription dose should cover 100% PTV and 95% PTV should receive 100% prescription dose. Total Lung: V20<23%, Dmean<13Gy, V5<50%. Spinal Cord: Dmax<40Gy. Heart: V30<40%, Dmean<25Gy. Esophagus: V40<5cc.

Treatment Implementation: Radiotherapy is implemented every day. Cone-beam CT should be utilized every day to minimize set-up error.

Follow-up: Patients should be follow-up every three months right after the completion of the final cycle of immunotherapy to 3 years after that. Then follow-up every half year is allowed to 5 years. After 5 years, follow-up every year is appropriate. In follow-up, chest CT and abdominal ultrasonography should be implemented. Cranial MRI should be performed every half year. Bone scan should be undertaken every year for all patients.

Inclusion Criteria:

1. 18-70 years old;
2. ECOG 0-1;
3. Adequate organ function to tolerate chemotherapy, immunotherapy and radiotherapy;
4. Small-cell lung cancer;
5. Limited stage confirmed by cranial MRI, chest CT, abdominal ultrasonograph, bone scan or cranial MRI and PET-CT;
6. Signature of inform consent.

Exclusion Criteria:

1. Younger than 18 years old or older than 70 years old;
2. ECOG>1;
3. Inadequate organ function to tolerate chemotherapy, immunotherapy and radiotherapy;
4. Non-small cell lung cancer and other neuroendocrine carcinoma including typical or atypical carcinoid, large-cell neuroendocrine carcinoma;
5. Extensive stage confirmed by cranial MRI, chest CT, abdominal ultrasonograph, bone scan or cranial MRI and PET-CT;
6. No signature of inform consent.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old;
* ECOG 0-1;
* Adequate organ function to tolerate chemotherapy, immunotherapy and radiotherapy;
* Small-cell lung cancer;
* Limited stage confirmed by cranial MRI, chest CT, abdominal ultrasonograph, bone scan or cranial MRI and PET-CT;
* Signature of inform consent.

Exclusion Criteria:

* Younger than 18 years old or older than 70 years old;
* ECOG>1;
* Inadequate organ function to tolerate chemotherapy, immunotherapy and radiotherapy;
* Non-small cell lung cancer and other neuroendocrine carcinoma including typical or atypical carcinoid, large-cell neuroendocrine carcinoma;
* Extensive stage confirmed by cranial MRI, chest CT, abdominal ultrasonograph, bone scan or cranial MRI and PET-CT;
* No signature of inform consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 1 to 2 years
  progression-free survival

SECONDARY OUTCOMES:
2-year progression-free survival rate | 2 year
  2-year progression-free survival rate
2-year overall survival rate | 2 year
  2-year overall survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provicial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No